CLINICAL TRIAL: NCT03690141
Title: A Phase 2 Non-randomized Open-label Study Examining the Effect of Tomivosertib (eFT508) in Patients With Advanced Castrate-resistant Prostate Cancer (CRPC)
Brief Title: An Open-label Study of the Effect of Tomivosertib (eFT508) in Patients With Advanced Castrate-resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early due to a lack of efficacy.
Sponsor: Effector Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eFT508-0009
Record Dates: First submitted 2018-09-10; First posted 2018-10-01 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Castrate-resistant Prostate Cancer (CRPC)
Keywords: Prostate Cancer; Castrate-resistant Prostate Cancer; CRPC; eFT508; eFT508-0009; tomivosertib
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tomivosertib

STUDY DESIGN:
Intervention Model Description: tomivosertib (eFT508) will be supplied as 100-mg capsules by the Sponsor. Capsules are packaged in 200-cc high-density polyethylene wide-mouth, round, white bottles, at either 100 or 150 units per bottle, induction sealed and capped with a 38-mm child-resistant closure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tomivosertib (eFT508) (Experimental): Tomivosertib (eFT508) is a novel small-molecule, investigational drug being developed by eFFECTOR Therapeutics, Inc. as an anticancer therapy. Tomivosertib (eFT508) down regulates AR and acts by inhibiting mitogen-activated protein kinase-interacting serine/threonine kinase-1 (MNK1) and MNK2.
  Interventions: Drug: eFT508

INTERVENTIONS:
Drug: eFT508 — This Phase 2 study examines the efficacy, safety, tolerability, and PK of tomivosertib (eFT508) in advanced CRPC patients who have documented PSA progression on treatment with apalutamide and/or abiraterone and/or enzalutamide and for whom no suitable curative therapy exists.
  Other Names: tomivosertib

SUMMARY:
This Phase 2 Open-label Study examines the efficacy, safety, tolerability, and pharmacokinetics (PK) of tomivosertib (eFT508) in Patients with advanced CRPC.

An Open-label Study Examining the Effect of tomivosertib (eFT508) in Patients with Advanced Castrate-resistant Prostate Cancer (CRPC)

DETAILED DESCRIPTION:
This Phase 2 study examines the efficacy, safety, tolerability, and pharmacokinetics (PK) of tomivosertib (eFT508) in advanced CRPC patients who have documented PSA progression on treatment with apalutamide and/or abiraterone and/or enzalutamide and for whom no suitable curative therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Histologically or cytologically confirmed (by clinical site) adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features.
* Ongoing androgen deprivation therapy with a GnRH analog or bilateral orchiectomy (surgical or medical castration).
* Serum testosterone ≤1.73 nmol/L (50 ng/dL) at screening.
* PSA progression on treatment with abiraterone and/or enzalutamide and/or apalutamide. PSA progression is defined by a minimum of 2 rising PSA levels with an interval of ≥1 week between each determination. PSA value at the screening visit should be ≥2 ng/mL. Patients may also have:

  * Soft tissue disease progression defined by iRECIST/RECIST 1.1
  * Bone disease
* Patients receiving bisphosphonate/receptor activator of nuclear factor kappa-Β ligand (RANKL) therapy must have been on stable doses for ≥ 4 weeks before the start of study therapy.
* Completion of all previous therapy for the treatment of cancer ≥4 weeks before the start of study therapy.
* All acute toxic effects of any prior anti-tumor therapy resolved to Grade ≤1 before the start of study therapy (with the exception of alopecia [Grade 1 or 2 permitted], neurotoxicity [Grade 1 or 2 permitted], or bone marrow parameters [Grade 1 or 2 permitted with exceptions as noted below]).
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) ≥1.0 x 109/L
  * Platelet count ≥75 x 109/L
  * Hemoglobin ≥80 g/L (8.0 g/dL or 4.9 mmol/L)
* Adequate hepatic function:

  * Serum alanine aminotransferase (ALT) ≤3 x upper limit of normal (ULN), ≤ 5 x ULN in the presence of liver metastases
  * Serum aspartate aminotransferase (AST) ≤3 x ULN, ≤5 x ULN in presence of liver metastases
  * Serum bilirubin ≤1.5 x ULN (unless due to Gilbert's syndrome or hemolysis ≤3 x ULN)
* Adequate renal function:

  -Serum creatinine ≤1.5 mg/dL and/or creatinine clearance ≥30 mL/min using Cockcroft Gault equation (Appendix 13.4)
* For male patients who can father a child and are having intercourse with females of childbearing potential, willingness to use a protocol-recommended method of contraception from the start of study therapy and for ≥30 days following the last dose of study medication or to abstain from sexual intercourse for at least this period of time, and willingness to refrain from sperm donation from the start of study therapy to ≥90 days following the last dose of study drug.
* Estimated life expectancy >12 weeks.
* Willingness to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests and biopsies, other study procedures, and study restrictions. Note: Psychological, social, familial, or geographical factors that might preclude adequate study participation should be considered.
* Evidence of a personally signed informed consent indicating that the patient is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, possible side effects, potential risks and discomforts, and other pertinent aspects of study participation.

Exclusion Criteria:

* History of another malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin; adequately treated, papillary, noninvasive bladder cancer; other adequately treated Stage 1 or 2 cancers currently in complete remission, or any other cancer that has been in complete remission for ≥2 years.
* Rapidly progressive, clinically unstable central nervous system malignancy. Note: Central nervous system imaging is only required in patients with known or suspected central nervous system malignancy.
* Significant cardiovascular disease, including myocardial infarction, arterial thromboembolism, or cerebrovascular thromboembolism within 6 months before the start of study therapy; symptomatic dysrhythmias or unstable dysrhythmias requiring medical therapy; unstable angina; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure; Grade ≥3 hypertension (diastolic blood pressure ≥100 mmHg or systolic blood pressure ≥160 mmHg), or history of congenital prolonged QT syndrome.
* Significant screening electrocardiogram (ECG) abnormalities, including unstable cardiac arrhythmia requiring medication, left bundle-branch block, 2nd-degree atrioventricular (AV) block type II, 3rd-degree AV block, Grade ≥2 bradycardia, or QTcF ≥470 msec.
* Symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable.
* Patients with gastrointestinal disorders likely to interfere with absorption of study medication.
* Major surgery within 4 weeks before the start of study therapy.
* Prior treatment with chemotherapy within 3 weeks or at least 4 half-lives, whichever is longer, before the start of study therapy.
* Prior therapy with any known inhibitor of MNK-1 or MNK-2.
* Treatment with 5-alpha reductase inhibitors within 4 weeks of enrollment.
* Prior flutamide treatment within 4 weeks before the start of study therapy and evidence of withdrawal response.
* Bicalutamide or nilutamide within 6 weeks before the start of study therapy and evidence of withdrawal response.
* Enzalutamide or abiraterone or apalutamid within 4 weeks before the start of study therapy.

  a. Steroids given in conjunction with abiraterone must be washed out for at least 2 weeks prior to Cycle 1 Day 1 unless the investigator chooses to maintain at a dose of ≤10 mg/day prednisone or equivalent.
* Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (eg, saw palmetto).
* Current use of immunosuppressive medication at the time of randomization, EXCEPT for the following:

  1. intranasal, inhaled, topical steroids, or local steroid injection (eg, intra-articular injection);
  2. Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent;
  3. Steroids as premedication for hypersensitivity reactions (eg, computed tomography [CT] scan premedication).
* Use of a potent inhibitor or inducer of cytochrome P450 (CYP) 3A4 within 7 days before the start of study therapy or expected requirement for use of a CYP3A4 inhibitor or inducer during study therapy (Appendix 13.5).
* Concurrent participation in another therapeutic clinical trial.
* Any illness, medical condition, organ system dysfunction, or social situation, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, adversely affect the patient's ability to cooperate and participate in the study, or compromise the interpretation of study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyon Gliech, MD, Study Director — Medpace, Inc.
Locations (10):
- United States (10):
  - Yale Cancer Center, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - Kimmel Center at Johns Hopkins, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - The Urology Group, Cincinnati, Ohio
  - Lancaster Urology, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2 study examined the efficacy, safety, tolerability, and pharmacokinetics (PK) of tomivosertib in advanced castrate-resistant prostate cancer (CRPC) patients who had documented prostate-specific antigen (PSA) progression on treatment with apalutamide, and/or abiraterone, and/or enzalutamide for whom no suitable curative therapy existed. Study initiation date is 27 November 2018. On 26 June 2019 the study was terminated due to lack of efficacy.
Groups:
- Tomivosertib (eFT508) 200 mg Twice Daily: Tomivosertib (eFT508) is a novel small-molecule, investigational drug being developed by eFFECTOR Therapeutics, Inc. as an anticancer therapy. Tomivosertib (eFT508) down regulates AR and acts by inhibiting mitogen-activated protein kinase-interacting serine/threonine kinase-1 (MNK1) and MNK2.
  tomivosertib (eFT508): This Phase 2 study examines the efficacy, safety, tolerability, and PK of tomivosertib (eFT508) in advanced CRPC patients who have documented PSA progression on treatment with apalutamide and/or abiraterone and/or enzalutamide and for whom no suitable curative therapy exists.
  Study drug was administered in 4-week (28-day) treatment cycles. Patients self-administered tomivosertib orally at 200 mg twice daily.
Period: Overall Study
Arm/Group | Tomivosertib (eFT508) 200 mg Twice Daily
Started | 16
Completed | 0
Not Completed | 16
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 4
Not completed — Disease progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | Tomivosertib (eFT508) 200 mg Twice Daily
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (11.47)
Age, Continuous [Median (Full Range); unit: years] | 67.5 [42 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 13
  Black or African American | 3
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Anti-tumor Response as Defined by a Patient Achieving Either of the Following Outcomes:
Description: * A ≥50% PSA decline from baseline at any time point after therapy and maintained for ≥4 weeks
  * Objective response according to iRECIST 1.1
Time Frame: 52 weeks
Population: A total of 16 participants were enrolled to receive tomivosertib 200 mg. These 16 participants make up the Safety Population (i.e. any participant whom received ≥1 dose of eFT508).
Measure: Count of Participants; unit: Participants
Arm/Group | Tomivosertib (eFT508) 200 mg Twice Daily
Number analyzed (Participants) | 16
Participants | 0

2. Secondary Outcome: PSA Progression-free Survival From Start of Study Therapy Until the Date PSA Progression is First Observed.
Description: PSA progression is defined as a ≥25% increase in PSA from nadir or baseline (and by ≥2 ng/mL) and requires confirmation ≥3 weeks later.
Time Frame: 52 weeks
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Tomivosertib (eFT508): Tomivosertib (eFT508) is a novel small-molecule, investigational drug being developed by eFFECTOR Therapeutics, Inc. as an anticancer therapy. Tomivosertib (eFT508) down regulates AR and acts by inhibiting mitogen-activated protein kinase-interacting serine/threonine kinase-1 (MNK1) and MNK2.
  tomivosertib (eFT508): This Phase 2 study examines the efficacy, safety, tolerability, and PK of tomivosertib (eFT508) in advanced CRPC patients who have documented PSA progression on treatment with apalutamide and/or abiraterone and/or enzalutamide and for whom no suitable curative therapy exists.
Arm/Group | Tomivosertib (eFT508)
Number analyzed (Participants) | 16
Weeks | 8.1 [4.1 to 31.1]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose through 30 days after the last dose of study medication, with a mean duration of study drug treatment of 11.5 weeks per participant. All-Cause Mortality was assessed through study completion, up to 52 weeks.
Description: An AE is defined as any untoward medical occurrence in a clinical investigation patient administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and/or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational medicinal product, whether or not related to the investigational medicinal product.
Arm/Group | Tomivosertib (eFT508) 200 mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 5/16
Serious Adverse Events (participants affected / at risk) | 7/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tomivosertib (eFT508) 200 mg Twice Daily (N=16)
Chest Pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Obstructive Nephropathy (Renal and urinary disorders) | 1 (1)
Urinary bladder rupture (Renal and urinary disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tomivosertib (eFT508) 200 mg Twice Daily (N=16)
nausea (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Edema peripheral (General disorders) | 2 (2)
Tremor (Nervous system disorders) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Aspartate aminotransferase increase (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Obstructive nephropathy (Renal and urinary disorders) | 1 (1)
Urinary bladder rupture (Renal and urinary disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or presentation of the results of this study may only be made in compliance with the provisions outlined in the executed Clinical Trial Agreement. Publication of scientific and clinical data will follow the recommendations of the International Committee of Medical Journal Editors, the Consolidated Standards of Reporting Trials group, and Good Publication Practice.

DOCUMENTS (2):
  • Study Protocol (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03690141/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT03690141/SAP_001.pdf